CLINICAL TRIAL: NCT03223038
Title: Pediatric International Nutrition Study - a Prospective, Multicenter Cohort Study of Nutritional Practices and Outcomes in Pediatric Intensive Care Units Around the World
Brief Title: Pediatric International Nutrition Study 2018
Acronym: PINS 2018
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Nilesh M. Mehta, Associate Professor of Anesthesia, Boston Children's Hospital
Other Study IDs: P00025098
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pediatric Critical Illness
Keywords: Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention - exposure is mechanical ventilation in PICU

SUMMARY:
This is a multi-site study of how nutrition is delivered to critically ill patients in pediatric intensive care units (PICUs) around the world. Each site will include mechanically ventilated children in their respective PICUs and record the details of what type and amount of nutrition was received. These details will be compared to goals designated by the clinicians caring for each patient. Data will be entered in a secure online remote data capture tool and managed by the lead researchers in Pediatric Critical Care Nutrition at Boston Children's Hospital, Nilesh Mehta, MD and Lori Bechard, PhD, RD. Data will be analyzed to better understand how different types and amounts of nutrition impact important PICU outcomes such as length of stay, ventilator time, incidence of infections, and mortality.

DETAILED DESCRIPTION:
Specific aim 1: To examine the impact of energy and protein adequacy on clinical outcomes.

Specific aim 2: To describe world-wide patterns of nutritional therapies in the PICU.environment: use of guidelines/use of adjuncts (acid suppression, motility, etc.)/glycemic control strategy/etc. To describe these practices in subgroups of: cardiac, surgical, medical, oncology/stem cell transplant patients in the PICU.

Specific aim 3: To examine enteral nutrition practices, including timing, route (gastric vs. post pyloric), adjuncts, and enteral nutrition (EN) intolerance definitions, in PICU patients worldwide Specific aim 4: To examine the current practices around parenteral nutrition prescription during the first week of critical illness in the PICU; time of initiation (early vs. late), rationale, threshold for initiation.

Primary predictor: nutritional adequacy (energy, protein) Secondary predictors: nutritional status, use of guidelines/site level indicators (location, staffing), use of adjuncts (acid suppression, motility, etc.), EN intolerance, subgroups (cardiac, surgical, medical, oncology/stem cell transplant), EN route/timing

ELIGIBILITY:
Inclusion Criteria:

* Sites with at least 8 PICU beds with the capacity to designate a site-specific clinician for data collection, preferably a clinician with an interest in nutrition or a dietitian, are eligible to participate.
* Patients 1 month to 18 years of age, admitted to the PICU and requiring mechanical ventilation with an anticipated length of PICU stay of 3 days or more.

Exclusion Criteria:

* Sites with < 8 PICU beds and/or no available clinician for data collection
* Subjects < 1 month or > 18 years, PICU length of stay < 3 days, not mechanically ventilated, receiving compassionate care only towards end of life, or enrolled in a nutrition intervention trial

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients 1 month to 18 years of age, admitted to the PICU and requiring mechanical ventilation with an anticipated length of PICU stay of 3 days or more.
Sampling Method: Non-Probability Sample
Enrollment: 1944 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
60 day mortality | 60 days
  incidence of mortality over 60 days following admission to PICU
incidence of hospital acquired infections | 60 days
  the number of infections (urinary tract, ventilator-associated, respiratory, or surgical site) that are acquired following PICU admission

SECONDARY OUTCOMES:
ventilator-free days | 28 days
  the number of days not requiring ventilator support during hospitalization
hospital length of stay | 60 days
  the number of days patient remains in the hospital following admission to the PICU
PICU length of stay | 60 days
  the number of days patient remains in the PICU following admission
weight status | 10 days
  weight-for-age Z-scores as determined by WHO standard growth criteria
growth status | 10 days
  height-for-age Z-scores as determined by WHO standard growth criteria
nutritional status | 10 days
  BMI or weight-for-height Z-scores as determined by WHO standard growth criteria
body composition in subgroup | 10 days
  % fat mass and % lean mass as assessed by bioelectrical impedance spectroscopy in approved subgroup
glycemic control | 10 days
  evaluation of clinically obtained maximum and minimum blood glucose values and use of insulin

CONTACTS AND LOCATIONS:
Overall Officials: Nilesh M Mehta, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Velazco CS, Zurakowski D, Fullerton BS, Bechard LJ, Jaksic T, Mehta NM. Nutrient delivery in mechanically ventilated surgical patients in the pediatric critical care unit. J Pediatr Surg. 2017 Jan;52(1):145-148. doi: 10.1016/j.jpedsurg.2016.10.041. Epub 2016 Oct 28. PMID 27856012
- [Background] Bechard LJ, Mehta NM. Nutritional Assessment Must be Prioritized for Critically Ill Children in the PICU. Crit Care Med. 2017 Apr;45(4):e464. doi: 10.1097/CCM.0000000000002220. No abstract available. PMID 28291114
- [Background] Albert BD, Zurakowski D, Bechard LJ, Priebe GP, Duggan CP, Heyland DK, Mehta NM. Enteral Nutrition and Acid-Suppressive Therapy in the PICU: Impact on the Risk of Ventilator-Associated Pneumonia. Pediatr Crit Care Med. 2016 Oct;17(10):924-929. doi: 10.1097/PCC.0000000000000915. PMID 27509362
- [Background] Bechard LJ, Duggan C, Touger-Decker R, Parrott JS, Rothpletz-Puglia P, Byham-Gray L, Heyland D, Mehta NM. Nutritional Status Based on Body Mass Index Is Associated With Morbidity and Mortality in Mechanically Ventilated Critically Ill Children in the PICU. Crit Care Med. 2016 Aug;44(8):1530-7. doi: 10.1097/CCM.0000000000001713. PMID 26985636
- [Background] Mehta NM, Bechard LJ, Zurakowski D, Duggan CP, Heyland DK. Adequate enteral protein intake is inversely associated with 60-d mortality in critically ill children: a multicenter, prospective, cohort study. Am J Clin Nutr. 2015 Jul;102(1):199-206. doi: 10.3945/ajcn.114.104893. Epub 2015 May 13. PMID 25971721
- [Background] Martinez EE, Bechard LJ, Mehta NM. Nutrition algorithms and bedside nutrient delivery practices in pediatric intensive care units: an international multicenter cohort study. Nutr Clin Pract. 2014 Jun;29(3):360-7. doi: 10.1177/0884533614530762. Epub 2014 Apr 16. PMID 24740498
- [Background] Mehta NM, Bechard LJ, Cahill N, Wang M, Day A, Duggan CP, Heyland DK. Nutritional practices and their relationship to clinical outcomes in critically ill children--an international multicenter cohort study*. Crit Care Med. 2012 Jul;40(7):2204-11. doi: 10.1097/CCM.0b013e31824e18a8. PMID 22564954
- [Derived] Bechard LJ, Staffa SJ, Zurakowski D, Mehta NM. Time to achieve delivery of nutrition targets is associated with clinical outcomes in critically ill children. Am J Clin Nutr. 2021 Nov 8;114(5):1859-1867. doi: 10.1093/ajcn/nqab244. PMID 34320161
- See also: Pediatric Critical Care Nutrition website — http://picunutrition.org